CLINICAL TRIAL: NCT04884451
Title: Evaluation of a Stage-Based Tailored, Nutrition Education Package for Childhood Obesity (ST-NEPCO) (7-12 Years Old)
Acronym: ST-NEPCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Nor Baizura Md. Yusop, Dr, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JKEUPM-2019-375
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Educational Materials (ST-NEPCO) During Nutrition Counselling for Obese Children

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive nutritional counselling from the researcher based on Stage-Based, Nutrition Education Package for Childhood Obesity (ST-NEPCO). Nutritional advice and educational tools will be provided according to participants' stages of change.
  Interventions: Behavioral: Lifestyle modification
- Control (No Intervention): Participants will receive counseling from dietitians based on the routine care for the management of childhood obesity.

INTERVENTIONS:
Behavioral: Lifestyle modification — Diet and physical activity modification and behavioral approach
  Arms: Intervention

SUMMARY:
A randomized controlled trial will be used to determine the effectiveness of ST-NEPCO. The study will involve obese children aged 7 to 11 years old. Participants will be assigned randomly to either the intervention or control group. The intervention group will receive counselling from the researcher based on ST-NEPCO, meanwhile the control group will receive counseling from dietitians based on the routine care for the management of childhood obesity. The study will be conducted for duration of 24 weeks. The individual counseling session will be held once a month for each participant during the weekend.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 11 years old
* Children classified as obese (>+2SD) based on BMI-for-age for 5 to 19 years old (WHO, 2007).

Exclusion Criteria:

* Children diagnosed with chronic asthma, diabetes mellitus, psychiatric disorders (e.g. schizophrenia, severe autism or mental retardation, or psychosis), or other serious medical conditions.
* Children receiving medications that can potentially promote weight gain or weight loss.
* Children participating in any weight management program

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-04-03 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
BMI-for-age z -score change | Change from baseline to week 24
  BMI-for-age z-score will be calculated using the WHO AnthroPlus software (http://www.who.int/growthref/tools/en) and the WHO 2007 growth reference will be used to determine the BMI-for-age z-score of participants (de Onis et al., 2007).

SECONDARY OUTCOMES:
Body composition (BMI, Lean Body Mass (LBM), Body Fat Mass (BFM) change | Change from baseline to week 24
  Body composition was measured using a body composition analyzer (InBody S10®; Biospace Co., Ltd., Seoul, Korea). This device uses multiple frequencies (1 kHz, 5 kHz, 50 kHz, 250 kHz, 500 kHz, and 1,000 kHz) of BIA technology and contains 8-point tactile electrodes that were attached to the left and right thumb, middle finger, and ankles. Subjects were in stand position; their arms and legs did not come into contact with each other, and they did not talk or move during the measurement, which lasted 2 minutes.
Waist and hip circumferences change | Change from baseline to week 24
  WC will be measured using a fibreglass tape (measuring tape SECA 201 SECA Vogel and Halke Gmbh & Co., Germany) at the highest point of the iliac crest at minimal respiration when the participant in a standing position. HC will be obtained at the widest area of hips, which is at the greatest protuberance of the buttocks. The 90th percentile values for WC for sex and age by Poh et al. (2011) will be used as cut-off values to identify respondents with abdominal obesity.
Energy and nutrient intakes [macronutrients, Saturated Fatty Acids (SFA), sugar and dietary fibre] change | Change from baseline to week 24
  Dietary intake will be obtained using three-day food record at baseline and every follow-up visits. Participants and parents/caregivers will be taught about portion size estimation and household measurement to fill in the three-day food record. Pictures from the Atlas of Food Exchanges and Portion Sizes (food album) (Suzana et al., 2002), a set of household measurement tools (glass, soup bowl, plate, cup, teaspoon and tablespoon) and food models will be used to guide parents/caregivers in estimating portion sizes.
Physical activity score change | Change from baseline to week 24
  Physical activity will be assessed using The Physical Activity Questionnaire for Older Children (PAQ-C) (Kowalski et al., 2004). Subjects will be classified into low, moderate and high physical activity categories with a mean total score ranging from 1.00 to 2.33, 2.34 to 3.66 and 3.67 to 5.00, respectively (Baharudin et al., 2014; Kowalski et al., 2004). Internal consistency (Cronbach's alpha) calculated from baseline was 0.73.
Stage of readiness to lose weight change | Change from baseline to week 24
  The measurement will be based on the scale for SOC (The S-Weight) to assess the readiness to lose weight for overweight and obese individual. It consists of five options that are mutually exclusive, among which participants have to choose in order to be allocated to one of the five SOC (Ceccarini, Borrello, Pietrabissa, Manzoni, & Castelnuovo, 2015).

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Putra Malaysia Teaching Hospital, Serdang, Selangor, Malaysia